CLINICAL TRIAL: NCT05473091
Title: Is There a Link Between Inflammation and Endocrinopathies in Turner Syndrome?
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, EVA FEIGERLOVA, Dr, Central Hospital, Nancy, France
Other Study IDs: 2021pi189
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group
  Interventions: Other: no intervention
- Control group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — retrospective analysis

SUMMARY:
Liver abnormalities are common in Turner syndrome. The physiopathology of these abnormalities is unknown for the moment but their potentially serious evolution requires additional explorations.

ELIGIBILITY:
Inclusion Criteria Experimental group:

* Turner syndrome

Inclusion Criteria Control group:

* healthy subjects

Ages: 18 Years to 56 Years | Sex: Female
Age Groups: Adult
Study Population: Retrospective analysis of data from patients followed in the Service of Endocrinology, Diabetology and Nutrition, University Hospital of Nancy
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
pro inflammatory score | 18 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHUR de Nancy, Nancy, France